CLINICAL TRIAL: NCT03839576
Title: Motor Signature, Falls Risk, and Home-Based Interventions in Older Adults With Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MOST106-2314-B-038-046
Record Dates: First submitted 2019-01-31; First posted 2019-02-15 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-01

CONDITIONS: Mild Cognitive Impairment; Fall
Keywords: gait; computerized cognitive training; falls; mild cognitive impairment; mobility; physical exercise; tai chi chuan
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A single-blinded, randomized controlled trial is designed to compare the effects of social interaction, computerized cognitive training, lower extremity strengthening, and tai chi chuan on improving cognitive functions and gait/mobility and reducing falls.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Computerized cognitive training (Experimental): The computerized cognitive training will take place at each participant's residence. Participants will be asked to practice at least 1 session a day for 6 months, and a session lasts for 60 minutes.
  Interventions: Behavioral: Computerized training
- Lower extremity strengthening (Experimental): This exercise will comprise stretching, muscle strengthening, and balance training at increasing difficulty levels, tailored and supervised by a physical therapist, and will take place at a subject's residence or in the neighborhood once a week for 6 months.
  Each session will last 60 min.
  Interventions: Behavioral: Exercise
- Tai chi chuan (Experimental): The 8-form Yang-style tai chi intervention will take place at a subject's residence or the neighborhood once a week for 6 months, and each session will last for 60 minutes.
  Interventions: Behavioral: Exercise
- Social interaction (No Intervention): Immediately after the baseline assessment, the care manager will visit the subject in this group once for comparability with the other two intervention groups.

INTERVENTIONS:
Behavioral: Exercise — Each session will last 60 min, consisting of 10 min of warm-up, 45 min of exercise, and a 5-min cool-down.
  Arms: Lower extremity strengthening; Tai chi chuan
Behavioral: Computerized training — Attention, memory, speed of processing, and executive functioning.
  Arms: Computerized cognitive training

SUMMARY:
A single-blinded, randomized controlled trial is designed to compare the effects of social interaction, computerized cognitive training, lower extremity strengthening, and tai chi chuan on improving cognitive functions and gait/mobility and reducing falls among 228 subjects with mild cognitive impairment, in which the influence of adherence to the intervention programs will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years old
* Had a fall at least 3 months prior to the baseline assessment
* Can ambulate independently
* Has mild cognitive impairment

Exclusion Criteria:

* Cannot ambulate independently and communicate with researchers
* Have a major unstable cardiopulmonary disease (e.g., ischemic chest pain, shortness of breath, recurrent syncopal episodes, orthopnea, paroxysmal nocturnal dyspnea, palpitations, or tachycardia)
* Have a contraindication to physical exercise (e.g., severe osteoarthritis or severe pulmonary hypertension)

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2023-01-24 (Estimated); Study Completion 2023-01-24 (Estimated)

PRIMARY OUTCOMES:
Mattis Dementia Rating Scale (MDRS) | 12 months
  The Mattis Dementia Rating Scale (MDRS) contains five cognitive domains of attention, initiation/perseveration, construction, conceptualization, and memory, which specifically assess concentration, verbal fluency, visuospatial skills, analogical reasoning, and short-term memory, with score ranges for these domains of 0~37, 0~37, 0~6, 0~39, and 0~25 points, respectively, and a total score range of 0~144 points.
modified Telephone Interview of Cognitive Status (TICS-M) | 12 months
  The modified Telephone Interview of Cognitive Status (TICS-M) consists of the date of the interview, age, phone number, immediate and delayed word list recall, counting backward, responsive naming, word opposites, and repetition, with a total score range of 0~50.
mobility | 12 months
  The timed up and go test requires subjects to rise from a standard chair, walk a distance of 3 m, turn, walk back to the chair, and sit down. The time to complete the timed up and go will be recorded.
balance | 12 months
  The Tinetti balance score ranges 0~26, with a higher score indicating a better balance ability.
falls | 12 months
  number of falls and multiple falls

SECONDARY OUTCOMES:
depressive symptoms | 12 months
  Depressive symptoms will be assessed using the 15-item Geriatric Depression Scale.
fear of falling | 12 months
  Activities-specific Balance Confidence (ABC) scale assesses an individual's confidence in performing 16 common daily tasks without losing balance, and total scores of the ABC scale are determined by the accumulated average of each item score and range between 0 and 100, with lower scores indicating greater balance confidence.
activity of daily living (ADL) | 12 months
  The activity of daily living (ADL) scale consists of seven basic ADLs (self-feeding, self-dressing, grooming, walking, getting in/out of bed, bathing, and controlling the bladder) and seven instrumental ADLs (using a telephone, transporting oneself, shopping, preparing meals, doing housework, taking medication, and managing one's money). These items are graded as 0 points (inability), 1 point (needs some help), or 2 points (no help needed). The ADL score ranges from 0 to 28 points, with a lower score indicating greater activity disability.

CONTACTS AND LOCATIONS:
Overall Officials: Mau-Roung Lin, Professor, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No